CLINICAL TRIAL: NCT04531215
Title: Ultrasound Guided Retrolaminar Versus Erector Spinae Plane Block for Postoperative Analgesia in Modified Radical Mastectomy
Brief Title: Ultrasound Guided Retrolaminar Versus Erector Spinae Plane Block for Postoperative Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, clinical professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6236
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided Retrolaminar Block (Active Comparator): ultrasound guided Retrolaminar Block (RLB) with 20 ml (0.5% Bupivacaine) plus 5 mic/ml Adrenaline (1:200,000) at the level of T4 of the surgical side.
  Interventions: Drug: ultrasound guided Retrolaminar Block
- ultrasound guided erector spinae (Active Comparator): ultrasound guided Erector Spinae Plane Block (ESPB) with 20 ml (0.5% Bupivacaine) plus 5 mic/ml Adrenaline (1:200,000) at the level of T4 of the surgical side.
  Interventions: Drug: ultrasound guided Erector Spinae Plane

INTERVENTIONS:
Drug: ultrasound guided Retrolaminar Block — ultrasound guided Retrolaminar Block (RLB) with 20 ml (0.5% Bupivacaine) plus 5 mic/ml Adrenaline (1:200,000) at the level of T4 of the surgical side
  Arms: ultrasound guided Retrolaminar Block
Drug: ultrasound guided Erector Spinae Plane — ultrasound guided Erector Spinae Plane Block (ESPB) with 20 ml (0.5% Bupivacaine) plus 5 mic/ml Adrenaline (1:200,000) at the level of T4 of the surgical side.
  Arms: ultrasound guided erector spinae

SUMMARY:
Thoracic epidural anesthesia (TEA) and paravertebral block (PVB) have been utilized to give perioperative regional anesthesia in the trunk. TEA is technically troublesome in some cases, and is associated with a danger of serious complications, such as epidural hematoma, nerve injury, and hypotension. PVB has the benefit of perception of the needle position using ultrasonography. However, PVB is also additionally connected with a danger of serious complications, such as pneumothorax, hypotension, or nerve injury. Newer approaches to deal with PVB have been the focal point of numerous techniques lately; these methodologies incorporate retrolaminar block (RLB) and erector spinae plane block (ESPB)

DETAILED DESCRIPTION:
Modified radical mastectomy is one of the commonly performed breast surgery. Postoperative pain following mastectomy should be minimized, as in a number of women it may chronically persist for months in the form of post-mastectomy pain syndrome.

Morphine administration for acute pain after mastectomy surgery has many side effects. Regional block techniques as para-vertebral block and thoracic epidural anesthesia have possible complications and technical difficulties.

The new alternative regional techniques such as erector spinae plane block and retrolaminar block are clinical trials for providing a safe and easy with good hemodynamic and recovery profile with adequate perioperative analgesia for a large section of patients undergoing mastectomy operation in order to reduce opioids consumption and subsequently avoid opioid-related adverse effects.

As percent of post-operative rescue analgesia is 16.7% and 60% for RLB group and ESPB group respectively. So, sample size is 46 patients (23 patients in each group). Sample was calculated using OPEN EPI program with confidence level 95% and power 80%.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* 21 - 64 years of age.
* American Society of Anesthesiologist physical status class I,II.
* Body Mass Index 25-35 kg/m2.
* Female patient undergoing elective unilateral modified radical mastectomy under general anesthesia.

Exclusion Criteria:

* Coagulation disorders or anticoagulant therapy.
* Known allergy to study drugs (Bupivacaine, Fentanyl)
* Infection at the injection site.
* Patients having chronic pain or on pain treatment.
* Advanced renal, respiratory, hepatic or cardiovascular disorders.
* Uncooperative patients.
* Duration of surgery > 3hours.
* Pregnant or lactating females.
* Metastasis.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Total fentanyl dose. | from induction to end of surgery
  The anesthesiologist will administer intravenous fentanyl 0.5 μg/kg when the heart rate or blood pressure of the patients increased >20% from basal measurements after exclusion of other causes.

SECONDARY OUTCOMES:
pain intensity by Visual Analogue Scale | at 30 minutes then at 2, 4, 8, 12, 18 and 24 hours post-operatively.
  • Static and dynamic pain scores (VAS) at 30 minutes, 2, 4, 8, 12, 18 and 24 hours post-operatively.
  pain intensity will be evaluated by Visual Analogue Scale (VAS). VAS is a 10 cm horizontal line labeled "no pain" at one end and "worst pain" imaginable on the other end. The patient will be asked to mark on this line where the intensity of the patient lies.
Time of requirement of rescue dose of Fentanyl. | up to 24hour postoperative
  Time of requirement of rescue dose of Fentanyl.
Total amount of postoperative Fentanyl | up to 24hour postoperative
  Total amount of Fentanyl consumed during the first 24 hours after surgery.
Post-operative nausea and vomiting | up to 24hour postoperative
  • Post-operative nausea and vomiting will be noticed, recorded using a categorical scoring system (0 = none, 1 = mild, 2 = moderate, 3 = severe) and treated, Ondansetron 4 mg IV will be administered in case of reported nausea and/or vomiting
Complications including hypotension MAP < 60, bradycardia HR < 60b/m, nausea, vomiting and allergic reactions. | up to 24hour postoperative
  Complications including hypotension MAP < 60, bradycardia HR < 60b/m, nausea, vomiting and allergic reactions.
Overall patient satisfaction | up to 24hour postoperative
  • Overall patient satisfaction at the end of the 24 hours post-operative using short assessment patient satisfaction scale (SAPS scale fully satisfied, neutral satisfied or unsatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Kamel, M.D, Study Chair — Zagazig University
Locations (1):
- Zagazig University, Faculty of medicine, Zagazig, Egypt